CLINICAL TRIAL: NCT03370835
Title: Randomized Open-Label Crossover Trial Comparing Tolerability of a Cardioselective Beta-Blocker (Metoprolol-Succinate-ER) and a Non-Cardioselective Beta-Blocker (Carvedilol) in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Tolerability of Metoprolol-Succinate-ER and Carvedilol in COPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Greater Los Angeles Healthcare System (U.S. Federal Agency)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0027
Record Dates: First submitted 2016-12-20; First posted 2017-12-12 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Asthma; Adverse Effect of Beta-adrenoreceptor Antagonists
Keywords: Beta-Blocker; Chronic Obstructive Pulmonary Disease; COPD; Cardioselective
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma | interventions — Metoprolol; Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1 (Experimental): Metoprolol-succinate-ER 25mg daily weeks 0-2, 50mg daily weeks 2-4, 100mg daily weeks 4-6, 200mg daily weeks 6-8, 100mg daily week 9, 50mg daily week 10
  Carvedilol 3.125mg twice daily weeks 10-12, 6.25mg twice daily weeks 12-14, 12.5mg twice daily weeks 14-16, 25mg twice daily weeks 16-18
  Interventions: Drug: Metoprolol succinate ER; Drug: Carvedilol
- Sequence 2 (Active Comparator): Carvedilol 3.125mg twice daily weeks 0-2, 6.25mg twice daily weeks 2-4, 12.5mg twice daily weeks 4-6, 25mg twice daily weeks 6-8, 12.5mg twice daily week 9, 6.25mg twice daily week 10
  Metoprolol-succinate-ER 25mg daily weeks 10-12, 50mg daily weeks 12-14, 100mg daily weeks 14-16, 200mg daily weeks 16-18
  Interventions: Drug: Metoprolol succinate ER; Drug: Carvedilol

INTERVENTIONS:
Drug: Metoprolol succinate ER — Cardioselective beta-blocker
Drug: Carvedilol — Non-cardioselective beta-blocker

SUMMARY:
Use of beta-blockers has proven beneficial in patients with hypertension, heart failure, and in people who have suffered a heart attack. The use in patients who have Chronic Obstructive Pulmonary Disease (COPD) and reactive airway disease, however, has been limited due to possible side effects such as worsening of lung function or increasing airway spasms and asthma attacks. The purpose of this study is to find out if patients with COPD can tolerate being on a beta-blocker at doses recommended for the treatment of heart disease conditions. This study also seeks to find out if a selective beta-1 receptor beta-blocker is better than a non-selective beta-blocker in patients with mild to moderate COPD.

ELIGIBILITY:
Inclusion Criteria:

* 40 years of age or older
* Mild to moderate COPD as defined by the American Thoracic Society
* Current treatment with a beta-blocker for either hypertension, myocardial infarction, or congestive heart failure.

Exclusion Criteria:

* Recent (within 30 days) COPD exacerbation or requirement for oral steroid therapy within the last 6 months
* Any history of ventilator support requirement for COPD
* Patients with asthma or reactive airway disease (RAD) defined as obstructive lung disease with a >15% improvement in FEV1 with beta-agonist therapy
* Relative or absolute contraindication to beta-blocker therapy
* Exposure to any investigational drugs within the previous 30 days
* Patients with any concurrent disease or condition, which in the judgment of the investigator would make the patient inappropriate for participation in the study were excluded from this study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2004-06; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Percent Change in FEV1 | 0, 4, 8, 14, 18 weeks

SECONDARY OUTCOMES:
Mean dose | 0-4, 4-8, 10-14, 14-18 weeks
  Mean dose of beta-blocker achieved during low (weeks 0-4 and 10-14) and high (weeks 4-8, 14-18) treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Freny V Mody, MD, Principal Investigator — VA Greater Los Angeles Healthcare System
Locations (1):
- VA West Los Angeles Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No